CLINICAL TRIAL: NCT00216294
Title: An Open-Label, Dose Escalation, Pilot Study to Assess the Safety and Efficacy of Subcutaneous RG1068 (Synthetic Human Secretin) in Patients With Obsessive Compulsive Disorder (OCD)
Brief Title: Safety Study of the Drug RG1068 in Patients With Obsessive Compulsive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Shekhar, Anantha M.D., Ph.D. (Individual); Repligen Corporation (Industry)
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0407-32; 4587029
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Obsessive Compulsive Disorder (OCD)
Keywords: Obsessive Compulsive Disorder; RG 1068 (Synthetic Human Secretin)
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Secretin

ARMS (2):
- Currently treated with SSRI (Experimental)
  Interventions: Drug: RG1068 (Synthetic Human Secretin)
- Not currently treated with SSRI (Experimental)
  Interventions: Drug: RG1068 (Synthetic Human Secretin)

INTERVENTIONS:
Drug: RG1068 (Synthetic Human Secretin)

SUMMARY:
The purpose of this study is to determine the safety and tolerability of RG1068 (Synthetic Human Secretin) when administered three times weekly to outpatients with obsessive compulsive disorder (OCD), to determine the impact of multiple subcutaneous injections of RG1068 on the symptoms of OCD, as measured by changes in clinical scales, and to evaluate the effect of RG1068 on OCD patients' anxiety, quality of life, and depression.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation pilot study. Prospective participants will initially undergo a blinded placebo challenge to assess his or her ability to self-administer drug. A total of sixteen subjects, will be enrolled in one of two study arms (eight subjects per group), depending on whether or not they are receiving concurrent treatment with a Selective Serotonin Reuptake Inhibitor (SSRI). The first 8 patients enrolled will receive subcutaneous injections of RG1068 at 10 µg/kg and will be divided between those receiving SSRI's and those not receiving SSRI's. Those not receiving SSRI treatment will further be divided between newly diagnosed, SSRI-naïve patients and patients who received SSRI's in the past but who have discontinued treatment for at least twelve weeks prior to enrollment. If there are no drug-related serious adverse events, an additional eight patients will be enrolled and receive RG1068 at 20 µg/kg. This group will also be divided between those receiving SSRI's and those not receiving SSRI's. Those not receiving SSRI treatment will be further divided in the same manner as before; newly diagnosed, SSRI-naïve patients, and patients who received SSRI's in the past but who have discontinued treatment for at least twelve weeks prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. outpatients with a primary DSM-IV diagnosis of OCD
2. age 18-40 years, inclusive
3. moderate to severe symptoms of OCD: a) YBOCS score of ≥24; b) CGI-Severity ≥4; c) significant disruption of daily activities (≥2 on item 1 or 6 of the YBOCS); d) disruption of employment/education function (≥2 on item 2 or 7 of the YBOCS)
4. if not on SSRI, must: a) have discontinued treatment with an SSRI at least 12 weeks prior to study Day 1; b) or be treatment naïve.
5. if on SSRI: a) must have residual symptoms despite a three month trial of an adequate dose of an SSRI drug; b) must currently be on an SSRI for at least 16 weeks and on a stable regimen for at least 8 weeks prior to Day 1.
6. Competent to give informed consent.

Exclusion Criteria:

1. moderate to severe depression (MADRS >25)
2. significant risk of suicidal behavior at screening
3. surgical lesion of anterior capsule (capsulotomy) or cingulate gyrus (cingulotomy)
4. co-morbid tics, Tourette syndrome, schizo-obsessive disorder, pure obsessive disorder or Axis II disorder
5. first degree relative with Tourette syndrome
6. pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections (PANDAS)
7. current cognitive behavioral psychotherapy
8. history of sensitivity to any of the ingredients in the study drug
9. Clinically significant abnormality in any screening laboratory results
10. Clinically significant organic disease (other than OCD), including cardiovascular, hepatic, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or extenuating circumstances that, in the opinion of the Investigator, would interfere with the performance or interpretability of, or put the patient at risk from, the study procedures
11. a current, active or ongoing DSM-IV Axis I psychiatric disorder other than anxiety disorders, major depression, dysthymia, and depression not otherwise specified (but including organic mental syndromes or disorders and dementia) as long as these are secondary diagnoses.
12. women who are pregnant, breastfeeding, or refuse to use adequate birth control
13. diagnosis of alcohol or substance abuse and/or dependence in the past 6 months
14. participating in an investigational drug study within 28 days of Day 1
15. concomitantly using any psychotropic medication other than SSRI or chloral hydrate for sleep
16. receiving treatment with a monoamine oxidase inhibitor within 2 weeks, a depot neuroleptic within 6 months, or a neuroleptic, anxiolytic, or antidepressant on a daily basis in the 2 weeks prior to Day 1.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-02; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Change in Yale-Brown Obsessive Compulsive Scale and
Clinical Global Impression of Change Scale

SECONDARY OUTCOMES:
Change in Hamilton Anxiety Scale,
Montgomery-Asberg Depressing Rating Scale, and
the Sickness Impact Profile

CONTACTS AND LOCATIONS:
Overall Officials: Anantha Shekhar, MD, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- LaRue Carter Hospital, Indianapolis, Indiana, United States